CLINICAL TRIAL: NCT06469593
Title: AID-BEYOND: Automated Insulin Delivery for Type 1 Diabetes - Beyond Glucose Metrics
Brief Title: Automated Insulin Delivery for Type 1 Diabetes - Beyond Glucose Metrics
Acronym: AID-BEYOND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Kirsten Nørgaard, Professor, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-23074743
Record Dates: First submitted 2024-06-11; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Closed-loop insulin pump; Automated insulin delivery; AID systems; Artificial pancreas; Type 1 Diabetes; T1D; Sleep; Cognition; Cardiovascular risk; Inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Inflammation

STUDY DESIGN:
Intervention Model Description: Randomized, open-label study comparing type-1 diabetes patients receiving usual treatment, with patients transitioning to AID systems
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adults with type 1 diabetes (intervention) (Experimental)
  Interventions: Device: Automated insuling delivery system
- Adults with type 1 diabetes (control) (No Intervention)
- Children with type 1 diabetes (intervention) (Experimental): Pediatric population of 7-17 years, stratified 1:1 to two groups of 7-11 and ≥12 years accordingly
  Interventions: Device: Automated insuling delivery system
- Children with type 1 diabetes (control) (No Intervention): Pediatric population of 7-17 years, stratified 1:1 to two groups of 7-11 and ≥12 years accordingly

INTERVENTIONS:
Device: Automated insuling delivery system — Closed-loop insulin pumps including MiniMed 780G, Tandom T2-slim x2 and YpsoCamAPS
  Other Names: Closed-loop insulin pumps
  Arms: Adults with type 1 diabetes (intervention); Children with type 1 diabetes (intervention)

SUMMARY:
The goal of this clinical trial is to determine if transitioning to automated insulin delivery (AID) systems, can improve objectively measured sleep quality and quantity and alleviate cardiovascular risk factors in both children and adults diagnosed with type 1 diabetes. The main questions it aims to answer are:

* Does the intervention improve sleep efficiency as measured by the HomeSleepTest, EEG based device, 4 months after initiation?
* Can the use of AID treatment alleviate cardiovascular risk measured by heart rate variability (HRV), blood pressure and inflammatory markers?
* Researchers will compare AID systems to usual treatment, including both multiple daily injections and sensor augmented pumps to see if the above benefits can be achieved with AID in comparison. Participants will be randomized 1:1 to either start AID treatment or to continue their usual care. The study will be open label.

Participants will, at baseline and after 4 months:

* Have taken blood and urine samples to measure metabolic and inflammatory parameters
* Perform digital cognitive testing using the CANTAB software
* Fill out questionnaires related to quality of life, fear of hypoglycemia, hypoglycemia awareness, eating habits and sleep quality
* Wear a blinded CGM for 10 days
* Monitor sleep at home using the HomeSleepTest for 3 consecutive nights
* Wear a Holter monitor for 24 hours to determine HRV parameters
* Measure blood pressure for 24 hours at 30 min intervals
* Wear an ActiGraph for 7 days to assess sleep and activity, supported by daily electronic sleep diaries

Participants randomized to AID treatment will receive education in the use of the systems.

Virtual follow-up visits are scheduled at week 1, 5 and 9 for both control and intervention groups during the study, following baseline examinations.

ELIGIBILITY:
Inclusion Criteria (Adults):

* Age ≥18 years
* Type 1 diabetes ≥3 years
* CGM or intermittently scanned CGM (isCGM) use ≥6 months
* Approval from the responsible health care provider (HCP) to start AID
* Specific AID system chosen ahead of screening after participant has been thoroughly informed

Inclusion Criteria (Children):

* Age 7-17 years
* Type 1 diabetes ≥6 months
* CGM or isCGM use ≥6 months
* Approval from the responsible HCP to start AID
* Specific AID system chosen ahead of screening after participant has been thoroughly informed

Exclusion Criteria:

* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during the study period or within 30 days prior to study start
* Use of commercial or open-source AID systems prior to study participation
* Daily use of paracetamol (acetaminophen)
* Breast-feeding, pregnancy or planning to become pregnant within 4 months
* Alcohol or drug abuse
* Severe cardiac disease
* Retinopathy contraindicating HbA1c <53 mmol/mol
* Other concomitant medical or psychological condition that, according to the investigator's assessment, makes the person unsuitable for study participation
* Lack of compliance with key study procedures at the discretion of the investigator

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in change from baseline to study end in sleep efficiency between the two groups. | Baseline and week 18
  Measured by HomeSleepTest for 3 consecutive days. Expressed in percentage.

SECONDARY OUTCOMES:
Total sleep duration | Baseline and week 18
  As measured by HomeSleepTest for 3 consequtive days. Expressed in minutes.
Time in sleep stages | Baseline and week 18
  As measured by HomeSleepTest for 3 consequtive days. Expressed in minutes.
Time in sleep stages | Baseline and week 18
  As measured by HomeSleepTest for 3 consequtive days. Expressed in percentages.
Sleep latency | Baseline and week 18
  As measured by HomeSleepTest and ActiGraph for 3 consequtive days.Expressed in minutes
Waking after sleep onset | Baseline and week 18
  As measured by HomeSleepTest and Actigraph for 3 consequtive days. Expressed in minutes
24-hour blood pressure | Baseline and week 18
  Measured using SpaceLabs Ontrak. Expressed in mmHg, SBP, DBP and MAP means and differences at day/nighttime. Presence of nighttime dipping (defined as MAP reduction of 10% or more). Difference in dat day- and nighttime defined as time asleep measured by HST.
Heart rate variability | Baseline and week 18
  Measured using Bittium Faros 180 holter monitors for 24 hours. Measured as standard deviation of NN intervals in milliseconds.
Heart rate variability | Baseline and week 18
  Measured using Bittium Faros 180 holter monitors for 24 hours. Measured as root mean square of successive RR interval differences (rMSSD) in milliseconds.
Heart rate variability | Baseline and week 18
  Measured using Bittium Faros 180 holter monitors for 24 hours. Measured as frequency-domain distribution absolute power in milliseconds squared.
Heart rate variability | Baseline and week 18
  Measured using Bittium Faros 180 holter monitors for 24 hours. Measured as frequency-domain distribution relative power in percentage.
Cognitive function | Baseline and week 18
  Measured using Cambridge Neuropsychological Test Automated Battery (CANTAB) with the Rapid Visual Information Processing test for both the adult and pediatric population.
Cognitive function | Baseline and week 18
  Measured using Cambridge Neuropsychological Test Automated Battery (CANTAB) with the Delayed Matching to Sample test for both the adult and pediatric population.
Cognitive function | Baseline and week 18
  Measured using Cambridge Neuropsychological Test Automated Battery (CANTAB) with the Spatial Working Memory test for the adult population only.
Cognitive function | Baseline and week 18
  Measured using Cambridge Neuropsychological Test Automated Battery (CANTAB) with the Stop Signal Task test for the adult population only.
Inflammatory markers | Baseline and week 18
  Defined in fold changes to expression of IL-1β, IL-6, IL-8, TNF-α, MCP-1, VEGF-α, CRP, ICAM-1, V-CAM-1, CRP. Assessed using multiplex ELISA analyses with MesoScale V-Plex and S-Plex plates.
Hypoglycaemia Fear Survey scores | Baseline and week 18
  Possible scores between 0-44, higher scores mean more fear of hypoglycemia.
Diabetes Distress Scale scores | Baseline and week 18
  Possible scores between 7-42, higher scores mean more diabetes distress.
Pittsburgh Sleep Quality Index scores | Baseline and week 18
  Measured for adults only. Possible scores between 0-21, higher scores means more severe sleep issues.
EuroQol 5-Domain scores | Baseline and week 18
  For adults the 5 Likert scale (5Q-5D-5L) will be used. For children the Young scale (5Q-5D-Y) scale will be used.
5-item World Health Organization Well-Being Index (WHO-5) scores | Baseline and week 18
  Possible scores between 0-100. Lower scores means worse well-being.
Sleep Screening Questionnaire Children and Adolescents (SSQ-CA) scores | Baseline and week 18
  Measured for children
Sleep efficiency | Baseline and week 18
  Measured in percentages, assessed using 7 days of ActiGraph data, supported by daily electronic sleep diaries.
Wake time after sleep onset | Baseline and week 18
  Measured in minutes, assessed using 7 days of ActiGraph data, supported by daily electronic sleep diaries.

OTHER OUTCOMES:
HbA1c | Baseline and week 18
Time with glucose values in range of 3.9 -10.0 mmol/L | Baseline and week 18
  Measured in percentage.
Time with glucose values < 3.9 mmol/l | Baseline and week 18
  Measured in percentage.
Time with glucose values < 3.0 mmol/l | Baseline and week 18
  Measured in percentage.
Time with glucose values > 10.0 mmol/l | Baseline and week 18
  Measured in percentage.
Time with glucose values > 13.9 mmol/l | Baseline and week 18
  Measured in percentage.
Sensor glucose | Baseline and week 18
  Measured as mmol/l with mean values and standard deviations
Glucose coefficient of variation | Baseline and week 18
  Measured in percentage
Time with rapid glucose change (> 1,5 mmol/l/15 min) | Baseline and week 18
  Measured in percentage.
Bodyweight | Baseline and week 18
  Measured in kilograms.
BMI standard deviation scores | Baseline and week 18
  Measured in the pediatric population.
Total daily insulin dose | Baseline and week 18
  Measured in IE and assessed by 2-week insulin pump data downloads
Total daily carbohydrate intake | Baseline and week 18
  Measured in grams and assessed by 2-week insulin pump data downloads
Hypoglycaemia awareness status | Baseline and week 18
  Assessed by the Gold questionaire. Possible scores between 1-7 with 7 being worst hypoglycemia awareness.
Hypoglycaemia awareness status | Baseline and week 18
  Assessed by the Clarke questionaire. Possible scores between 0-7 with 7 being worst hypoglycemia awareness.
Hypoglycaemia awareness status | Baseline and week 18
  Assessed by the Pedersen-Bjergaard questionaire. Possible outcomes are "Aware", "Impaired" and "Unaware".
Energy expenditure | Baseline and week 18
  Measured in kcal and assessed with 7 days of ActiGraph data.
Physical activity level | Baseline and week 18
  Categorized as sedentary, light and moderate-to-vigorous levels, assessed with 7 days of ActiGraph data.
Number of severe hypoglycaemia events | Baseline and week 18
  Expressed in diffence in number of events from baseline to end. Defined as cognitive impairment requiring external assistance for recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Nørgaard, MD, Prof., Principal Investigator — Steno Diabetes Center Copenhagen; Kurt Kristensen, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (3):
- Denmark (3):
  - Steno Diabetes Center Copenhagen, Herlev, Greater Copenhagen
  - Steno Diabetes Center Aarhus, Aarhus
  - Diagnostisk Center, Regionshospitalet Silkeborg, Silkeborg

IPD SHARING:
Plan to Share IPD: No